CLINICAL TRIAL: NCT06267781
Title: Biomarkers of Disease PROgression and Myeloid Profiling in Patients With Relapsing Remitting Multiple Sclerosis Treated With Autologous Hematopoietic Stem Cell TRANSPLANTation and Second Line Therapies.
Brief Title: RRMS: Disease PROgression and Myeloid Profiling After Bone Marrow TRANSPLANTation and Second Line Therapies
Acronym: TRANSPLANTPRO
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, Professor, IRCCS San Raffaele
Other Study IDs: TRANSPLANT-PRO
Record Dates: First submitted 2024-01-30; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will collect the following sample from enrolled patients with RRMS:
  -Peripheral blood in Ethylenediamine tetraacetic acid (EDTA) at baseline and at 3, 6, 12 and 24 months after the treatment's initiation.
  In patients treated with aHSCT we will collect also a blood sample obtained after the stem cells mobilization (collected the same day of stem cells apheresis) and, when available, advanced material from autologous graft infusion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- aHSCT: n.10 patients with RRMS referred for pharmacological treatment with myeloablative autologous hematopoietic stem cell transplantation (aHSCT) according to clinical practice following the Italian pharmacological regulatory agency (AIFA) criteria and guidelines and recommendations from the European Society for Blood and Marrow Transplantation (EBMT) Autoimmune Diseases Working Party (ADWP) and the Joint Accreditation Committee of EBMT and ISCT (JACIE)
- BCDT: n.10 patients with RRMS referred for pharmacological treatment with anti-CD20 monoclonal antibody (ocrelizumab or ofatumumab - B cell depleting therapies) according to clinical practice following the Italian pharmacological regulatory agency (AIFA) criteria.
- LEM: n.10 patients with RRMS referred for pharmacological treatment with anti-CD52 monoclonal antibody (alemtuzumab) according to clinical practice following the Italian pharmacological regulatory agency (AIFA) criteria.

SUMMARY:
To study whether highly effective therapies can halt disease progression in people with multiple sclerosis by modulating the peripheral myeloid landscape.

DETAILED DESCRIPTION:
Due to the limited availability of treatment in progressive multiple sclerosis (PMS), an in-depth analysis to better understand (1) the effect of disease-modifying therapies (DMTs) in preventing transition to secondary PMS (SPMS) and (2) the progression-related pathogenetic mechanisms, is essential. This could contribute to change the MS therapeutic perspective halting the progression independent of relapse activity putative processes, beside the prevention of relapse-associated worsening. Myeloablative autologous haematopoietic stem cell transplantation (aHSCT) in relapsing remitting multiple sclerosis (RRMS), differently from other widely used highly effective DMTs such as ocrelizumab and alemtuzumab, could modulate the myeloid activity inducing - after the depletion induced by conditioning regimen - a homeostatic expansion and enhanced immune regulation of monocytes/macrophages and dendritic cells. Currently used DMTs do not primarily target microglia/macrophage-mediated inflammation, and the effect on the abovementioned immune population could account for the advantage of aHSCT, compared to ocrelizumab and alemtuzumab, on progression free survival (PFS). Indeed, alemtuzumab and ocrelizumab achieve a long-term PFS lower than aHSCT. The results of such analyses could guide clinical decisions that will have a long-term impact, given the chronicity of the diseases, the duration of therapies, and the long-lasting effects of some treatments.

Given this premise, by evaluating n.10 consecutively recruited patients with RRMS treated with myeloablative aHSCT in comparison with patients (n.10 per group) treated with anti-cluster of differentiation (CD) 52 monoclonal antibody (alemtuzumab) and anti-CD20 monoclonal antibody (ocrelizumab or ofatumumab), the aims of this longitudinal study are the following:

Aim 1: To evaluate the impact of the studied treatments (myeloablative aHSCT, alemtuzumab and ocrelizumab/ofatumumab) on biomarkers of disease progression in MS. Since to clinically evaluate conversion to SPMS a long follow-up is required, the evaluation of progression's surrogate biomarkers (clinical, neuroradiological and biological) will allow a better and faster identification of the disease course.

Aim 2: To characterize the myeloid compartments' longitudinal changes induced by each treatment (aHSCT, alemtuzumab and ocrelizumab/ofatumumab) in the enrolled patients.

Aim 3: To explore a correlation between characteristics of the myeloid profile and surrogate endpoints of disease progression, assessing whether the treatment-induced homeostatic expansion and enhanced immune regulation of the myeloid compartment are related to surrogate endpoints of progression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Signed written informed consent;
* A diagnosis of RRMS according to the 2017 Revisions of the McDonald Criteria;
* High clinical and magnetic resonance imaging (MRI) inflammatory disease activity (at least 2 clinical relapses, or one clinical relapse with gadolinium (Gd)- enhancing or new T2 MRI lesions at a separate time point, in the previous 12 months)
* Patients referred for pharmacological treatment with aHSCT, alemtuzumab or ocrelizumab /ofatumumab, according to clinical practice following the Italian pharmacological regulatory agency (AIFA) criteria and guidelines and recommendations from the European Society for Blood and Marrow Transplantation (EBMT) Autoimmune Diseases Working Party (ADWP) and the Joint Accreditation Committee of EBMT and ISCT (JACIE);

Exclusion Criteria:

* Diagnosis of PPMS or SPMS according to the 2017 McDonald criteria
* Known intolerances/allergies to the active substance or the excipients contained in the DMT and/or contraindications according to product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 male or female prospective patients with RRMS who, from clinical practice, may be referred for treatment with aHSCT, alemtuzumab or ocrelizumab/ofatumumab will be recruited. Treatment choice will be independent of participation in the study and should not be initiated with the aim of including the patient in the study. All patients will be required to sign an informed consent before the collection of data and biological material.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2027-09-02 (Estimated); Study Completion 2027-09-02 (Estimated)

PRIMARY OUTCOMES:
Number of fading/disappearing paramagnetic rim lesions (PRLs) | 2 years (baseline and at 6, 12 and 24 months after study treatment )
  Evolution of the paramagnetic rim lesions (PRLs), main biomarker of progression, evaluated longitudinally (proportion of stable vs. fading/disappearing PRLs in each group of patients)

SECONDARY OUTCOMES:
Surrogate biomarkers of disease progression (MSFC) | 2 years (baseline and at 6, 12 and 24 months after study treatment)
  Changes in multiple sclerosis functional composite score (MSFC) evaluated longitudinally
Surrogate biomarkers of disease progression (sNfL) | 2 years (baseline and at 6, 12 and 24 months after study treatment)
  Changes in serum neurofilament light chain (sNfL) evaluated longitudinally
Surrogate biomarkers of disease progression (RNFL) | 2 years (baseline and at 6, 12 and 24 months after study treatment)
  Changes in retinal nerve fibre layer (RNFL) thickness evaluated longitudinally
Surrogate biomarkers of disease progression (cortical lesions) | 2 years (baseline and at 6, 12 and 24 months after study treatment)
  Number of new cortical lesions
Surrogate biomarkers of disease progression (atrophy) | 2 years (baseline and at 6, 12 and 24 months after study treatment)
  Changes of brain volumes evaluated longitudinally
Changes in myeloid landscape | 2 years (baseline and at 3, 6, 12 and 24 months after study treatment)
  Peripheral blood myeloid line subpopulations changes induced by each therapy studied by cytofluorometric analysis

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Filippi, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT06267781/Prot_SAP_000.pdf